CLINICAL TRIAL: NCT00752128
Title: RESOLUTE International Registry: Evaluation of the Resolute Zotarolimus-Eluting Stent System in a 'Real-World' Patient Population
Acronym: R-Int
Status: Completed | Type: Observational
Sponsor: Medtronic Vascular (Industry)
Collaborators: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Other Study IDs: IP091
Record Dates: First submitted 2008-09-12; First posted 2008-09-15 (Estimated); Results first posted 2011-12-06 (Estimated); Last update posted 2013-04-25 (Estimated); Status verified 2013-04

CONDITIONS: Coronary Artery Disease; Cardiovascular Diseases
Keywords: Drug Eluting Stent; Interventional Cardiology; Percutaneous Coronary Intervention
MeSH Terms: conditions — Coronary Artery Disease; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Endeavor Resolute Zotarolimus-Eluting Coronary Stent System — Stent implantation

SUMMARY:
The primary objective of the RESOLUTE international registry is to document the safety and overall clinical performance of the Resolute Zotarolimus-Eluting Coronary Stent System in a 'real-world' patient population requiring stent implantation.

DETAILED DESCRIPTION:
As part of the broader clinical program of the Resolute stent, the RESOLUTE International registry will expand the experience and understanding of the device performance in a 'real-world' setting. The registry intends to enroll patients from a large number of centers under commercial usage conditions, with the aim to reflect 'real-world' usage as much as possible.

ELIGIBILITY:
Inclusion Criteria:

* Minimum legal age (18)
* Acceptable candidate for treatment with a drug-eluting stent in accordance with applicable guidelines
* Patient has consented to participate and authorized in writing the collection and release of medical information
* Elective use of the Endeavor Resolute stent

Exclusion Criteria:

* Pregnancy
* High probability of non-adherence to the follow-up requirements (due to social, psychological or medical reasons)
* Currently participating in another trial preventing routine hospital treatment
* Previous enrollment in the RESOLUTE International registry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patients eligible for drug-eluting stent implantation with the elective use of the Endeavor Resolute stent in one or more target lesions are candidates to be enrolled
Sampling Method: Non-Probability Sample
Enrollment: 2349 (Actual)
Dates: Start 2008-08; Primary Completion 2010-10 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Franz-Josef Neumann, MD, Principal Investigator — Heart Center Bad Krozingen, Germany; Petr Widimský, MD, Principal Investigator — University Hospital Kralovské Vinohrady, Czech Republic; Jorge A. Belardi, MD, Principal Investigator — Instituto Cardiovascular de Buenos Aires, Argentina
Locations (1):
- Heart Center Bad Krozingen, Bad Krozingen, Germany

REFERENCES:
- [Derived] Silber S, Kirtane AJ, Belardi JA, Liu M, Brar S, Rothman M, Windecker S. Lack of association between dual antiplatelet therapy use and stent thrombosis between 1 and 12 months following resolute zotarolimus-eluting stent implantation. Eur Heart J. 2014 Aug 1;35(29):1949-56. doi: 10.1093/eurheartj/ehu026. Epub 2014 Feb 7. PMID 24510638
- [Derived] Richardt G, Leschke M, Abdel-Wahab M, Toelg R, El-Mawardy M, Serruys PW, Silber S, Windecker S, Belardi JA, Neumann FJ, Widimsky P; RESOLUTE All Comers; RESOLUTE International Investigators. Clinical outcomes of the Resolute zotarolimus-eluting stent in patients with in-stent restenosis: 2-year results from a pooled analysis. JACC Cardiovasc Interv. 2013 Sep;6(9):905-13. doi: 10.1016/j.jcin.2013.04.017. Epub 2013 Aug 14. PMID 23954063
- [Derived] Silber S, Serruys PW, Leon MB, Meredith IT, Windecker S, Neumann FJ, Belardi J, Widimsky P, Massaro J, Novack V, Yeung AC, Saito S, Mauri L. Clinical outcome of patients with and without diabetes mellitus after percutaneous coronary intervention with the resolute zotarolimus-eluting stent: 2-year results from the prospectively pooled analysis of the international global RESOLUTE program. JACC Cardiovasc Interv. 2013 Apr;6(4):357-68. doi: 10.1016/j.jcin.2012.11.006. Epub 2013 Mar 20. PMID 23523454
- [Derived] Farooq V, Vranckx P, Mauri L, Cutlip DE, Belardi J, Silber S, Widimsky P, Leon M, Windecker S, Meredith I, Negoita M, van Leeuwen F, Neumann FJ, Yeung AC, Garcia-Garcia HM, Serruys PW. Impact of overlapping newer generation drug-eluting stents on clinical and angiographic outcomes: pooled analysis of five trials from the international Global RESOLUTE Program. Heart. 2013 May;99(9):626-33. doi: 10.1136/heartjnl-2012-303368. Epub 2013 Mar 6. PMID 23468513

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Start recruitment: August 28, 2008 > End recruitment: March 19, 2009
Period: Overall Study
Arm/Group | Resolute Drug-Eluting Stent
Started | 2349
Completed | 2345
Not Completed | 4
Not completed — Withdrawal by Subject | 4

BASELINE CHARACTERISTICS:
Arm/Group | Resolute Drug-Eluting Stent
Number analyzed (Participants) | 2349
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1260
  >=65 years | 1089
Age Continuous [Mean (Standard Deviation); unit: years] | 63.5 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 521
  Male | 1828
Region of Enrollment [Number; unit: participants]
  Europe | 2118
  India | 174
  Argentina | 17
  South Africa | 40

OUTCOME MEASURES:

1. Primary Outcome: Composite Endpoint of Cardiac Death and Myocardial Infarction (Not Clearly Attributable to a Non-target Vessel)
Time Frame: 12 Months
Population: Analysis per intention to treat
Measure: Number; unit: percentage of participants
Groups:
- Cardiac Death or Target Vessel MI: Percentage of participants that had either Cardiac Death or Myocardial Infarction (not clearly attributable to a non-target vessel)
Arm/Group | Cardiac Death or Target Vessel MI
Number analyzed (Participants) | 2334
percentage of participants | 4.2

2. Secondary Outcome: Overall Stent Thrombosis, Defined as Definite and Probable Stent Thrombosis, According to the Academic Research Consortium (ARC) Definition
Time Frame: 12 Months
Population: Intention to treat
Measure: Number; unit: percentage of participants
Groups:
- Overall Stent Thrombosis (Definite and Probable-ARC): Overall stent thrombosis, defined as definite and probable stent thrombosis, according to the Academic Research Consortium (ARC) definition
Arm/Group | Overall Stent Thrombosis (Definite and Probable-ARC)
Number analyzed (Participants) | 2334
percentage of participants | 0.9

ADVERSE EVENTS:
Arm/Group | Resolute Drug-Eluting Stent
Serious Adverse Events (participants affected / at risk) | 33/2334
Other Adverse Events (participants affected / at risk) | 0/2334
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Resolute Drug-Eluting Stent (N=2334)
Cardiac Death (Cardiac disorders) | 33 (2334)

LIMITATIONS AND CAVEATS:
The data collection in this registry was limited to the collection of MACE (death, myocardial infarction (Q- and non-Q-wave), emergent cardiac bypass surgery and TLR) and stent thrombosis events.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other